CLINICAL TRIAL: NCT07013812
Title: Role of Tranexamic Acid in Control of Intraoperative Blood Loss in Women Undergoing Elective Cesarean Section
Brief Title: Tranexamic Acid to Reduce Blood Loss in Women Having Planned Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Combined Military Hospital Multan (Other)
Responsible Party: Principal Investigator, Hania Wahid, Principal Investigator, Combined Military Hospital Multan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U1111-1323-6469
Record Dates: First submitted 2025-05-30; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Cesarean Section; Blood Loss During Surgery
Keywords: Tranexamic acid; Elective Cesarean Section; Intraoperative blood loss
MeSH Terms: interventions — Tranexamic Acid; Glucose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Tranexamic Acid (Experimental): Patients received 1 g (10 ml) of tranexamic acid diluted in 20 mL of glucose 5%. Fifteen minutes before the surgery, the solution was injected intravenously slowly over a period of 5 minutes.
  Interventions: Drug: Tranexamic Acid (IV); Drug: Dextrose 5% (D5W)
- Intravenous 5% Dextrose (Placebo Comparator): Patients in this group received 30 mL of glucose 5%. Fifteen minutes before the surgery, the solution was injected intravenously slowly over a period of 5 minutes.
  Interventions: Drug: Dextrose 5% (D5W)

INTERVENTIONS:
Drug: Tranexamic Acid (IV) — One gram (10 ml) intravenous injection
  Other Names: TXA; Cyklokapron; Lysteda; Transamin.
  Arms: Intravenous Tranexamic Acid
Drug: Dextrose 5% (D5W) — 5% dextrose water intravenously

SUMMARY:
This clinical trial was done to find out if tranexamic acid (TXA) can safely reduce the amount of blood loss during cesarean (C-section) deliveries. Heavy bleeding is a major risk during childbirth, especially in C-sections, and can be life-threatening.

The main question this study wanted to answer was:

Does giving tranexamic acid before surgery reduce the amount of blood lost during a planned C-section?

In this study, 68 women who were scheduled for elective (planned) C-section deliveries were randomly assigned to receive either tranexamic acid or a placebo (a look-alike substance with no medicine in it) before surgery. The medication was given by slow injection just 15 minutes before the operation.

All surgeries followed the same procedure and were done by experienced obstetric surgeons. The amount of blood lost during surgery was carefully measured and compared between the two groups.

The goal was to find a simple and safe way to lower the risk of blood loss and its complications during C-sections, improving outcomes for mothers.

ELIGIBILITY:
Inclusion Criteria:

* Women age 20-45 years
* at 37-40 weeks of gestation (on LMP)
* Planned to undergo cesarean section under spinal anesthesia

Exclusion Criteria:

* Women with previous history of thromboembolic events
* Allergy to tranexamic acid
* Women with morbidly adherent placenta (on antenatal USG)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Blood Loss | During the elective cesarean section procedure
  Intraoperative blood loss (ml) was measured by taking weight difference of the dressings and towels before and after the operation plus blood added to the fluid volume inside the suction apparatus.

CONTACTS AND LOCATIONS:
Overall Officials: Nidda Y Professor, FCPS, Study Chair — Combined Military Hospital Multan
Locations (1):
- Combined Military Hospital, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abu-Zaid A, Baradwan S, Badghish E, AlSghan R, Ghazi A, Albouq B, Khadawardi K, AlNaim NF, AlNaim LF, Fodaneel M, AbuAlsaud FS, Jamjoom MZ, Almubarki AA, Alsehaimi SO, Alabdrabalamir S, Alomar O, Al-Badawi IA, Salem H. Prophylactic tranexamic acid to reduce blood loss and related morbidities during hysterectomy: a systematic review and meta-analysis of randomized controlled trials. Obstet Gynecol Sci. 2022 Sep;65(5):406-419. doi: 10.5468/ogs.22115. Epub 2022 Jul 28. PMID 35896179
- [Background] Shalaby MA, Maged AM, Al-Asmar A, El Mahy M, Al-Mohamady M, Rund NMA. Safety and efficacy of preoperative tranexamic acid in reducing intraoperative and postoperative blood loss in high-risk women undergoing cesarean delivery: a randomized controlled trial. BMC Pregnancy Childbirth. 2022 Mar 14;22(1):201. doi: 10.1186/s12884-022-04530-4. PMID 35287618